CLINICAL TRIAL: NCT01453725
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study of the Effect of Golimumab Administered Subcutaneously in Subjects With Active Axial Spondyloarthritis (Protocol No. P07642, Also Known as MK-8259-006-02).
Brief Title: Effect of Golimumab in Participants With Active Axial Spondyloarthritis (P07642, MK-8259-006)
Acronym: GO-AHEAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P07642; MK-8259-006 (Other: Merck Study Number); 2011-000311-34 (EudraCT Number)
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Results first posted 2014-12-18 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-01

CONDITIONS: Spondylitis, Ankylosing
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — golimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Golimumab→Golimumab (Experimental): In Part 1, participants receive golimumab 50 mg, administered subcutaneously (SC) every 4 weeks for up to 12 weeks (16 weeks of treatment). In Part 2, participants receive golimumab 50 mg, administered SC every 4 weeks for up to 28 weeks (32 weeks of treatment). (Combined total of up to 48 weeks treatment with golimumab.)
  Interventions: Biological: Golimumab
- Placebo→Golimumab (Placebo Comparator): In Part 1, participants receive placebo, administered SC every 4 weeks for up to 12 weeks (16 weeks of treatment). In Part 2, participants receive golimumab 50 mg, administered SC every 4 weeks for up to 28 weeks (32 weeks of treatment). (Combined total of up to 32 weeks treatment with golimumab.)
  Interventions: Biological: Golimumab; Biological: Placebo

INTERVENTIONS:
Biological: Golimumab — Golimumab 50 mg SC injection every 4 weeks
Biological: Placebo — Placebo SC injection every 4 weeks
  Arms: Placebo→Golimumab

SUMMARY:
This two-part study was to evaluate the effect of golimumab (SCH 900259, MK-8259) in participants with active axial spondyloarthritis (axial SpA). In Part 1, participants were to receive golimumab 50 mg or matching placebo subcutaneous injections on Day 1 (Baseline) and at Weeks 4, 8, and 12. During Part 1 of the study, participants were to not know the identity of the injection. In the Part 2 extension, all participants were to receive golimumab 50 mg subcutaneous injections beginning on Week 16 and then every 4 weeks up to Week 48. In Part 2, the participants were to be told they were receiving active study drug. The primary hypothesis of this study was that treatment with golimumab 50 mg every 4 weeks is superior to placebo as measured by the proportion of participants achieving an Assessment in Ankylosing Spondylitis (ASAS) 20 response at Week 16.

ELIGIBILITY:
Inclusion Criteria:

* Active axial spondyloarthritis with disease duration ≤5 years, and chronic back pain of ≥3 month duration
* Have either an inadequate response to 30 days of optimal daily doses of at least one non-steroidal anti-inflammatory drug (NSAID) or must be unable to receive a full 30 day maximal NSAID therapy because of intolerance, toxicity or contraindications to NSAIDs
* Females of child-bearing potential must use contraception
* No history of untreated latent or active tuberculosis

Exclusion Criteria:

* Fulfillment of modified New York criteria for ankylosing spondylitis
* Has ever received tumor necrosis factor (TNF)-α targeted therapy or any biological agents
* Any systemic inflammatory condition other than spondyloarthritis
* Serious infection within 2 months
* Any known malignancy or a history of malignancy within the previous 5 years
* Has or had a substance abuse (drug or alcohol) problem within the previous 2 years

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 198 (Actual)
Dates: Start 2012-02-13 (Actual); Primary Completion 2014-03-11 (Actual); Study Completion 2015-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Sieper J, van der Heijde D, Dougados M, Maksymowych WP, Scott BB, Boice JA, Berd Y, Bergman G, Curtis S, Tzontcheva A, Huyck S, Weng HH. A randomized, double-blind, placebo-controlled, sixteen-week study of subcutaneous golimumab in patients with active nonradiographic axial spondyloarthritis. Arthritis Rheumatol. 2015 Oct;67(10):2702-12. doi: 10.1002/art.39257. PMID 26139307
- [Derived] van der Heijde D, Dougados M, Maksymowych WP, Bergman G, Curtis SP, Tzontcheva A, Huyck S, Philip G, Sieper J. Long-term tolerability and efficacy of golimumab in active non-radiographic axial spondyloarthritis: results from open-label extension. Rheumatology (Oxford). 2022 Feb 2;61(2):617-627. doi: 10.1093/rheumatology/keab346. PMID 33878154
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P07642&kw=8259-006&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: These data are for Parts 1 and 2 of the study.
Period: Overall Study
Arm/Group | Golimumab→Golimumab | Placebo→Golimumab
Started | 98 | 100
Completed | 85 | 89
Not Completed | 13 | 11
Not completed — Adverse Event | 3 | 3
Not completed — Lost to Follow-up | 4 | 0
Not completed — Non-compliance With Protocol | 1 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Pregnancy Wish | 0 | 2
Not completed — Pregnancy | 1 | 0
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population consisted of all randomized participants.
Groups:
- Golimumab→Golimumab: In Part 1, participants receive golimumab 50 mg, administered SC every 4 weeks for up to 12 weeks (16 weeks of treatment). In Part 2, participants receive golimumab 50 mg, administered SC every 4 weeks for up to 28 weeks (32 weeks of treatment). (Combined total of up to 48 weeks treatment with golimumab.)
- Total: Total of all reporting groups
Arm/Group | Golimumab→Golimumab | Placebo→Golimumab | Total
Number analyzed (Participants) | 98 | 100 | 198
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.7 (7.1) | 31.7 (7.2) | 31.2 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 48 | 85
  Male | 61 | 52 | 113

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an Assessment in Ankylosing Spondylitis (ASAS) 20 Response at Week 16
Description: The ASAS consists of 4 domains: participant global assessment, total back pain, function (Bath Ankylosing Spondylitis Functional Index [BASFI]), and inflammation (mean of questions 5 and 6 of Bath Ankylosing Spondylitis Disease Activity Index [BASDAI]). Each domain is measured on a 100-mm visual analog scale (VAS) from 0 mm=the very best situation to 100 mm=the very worst situation, with a higher score indicating more severe impairment. ASAS 20 is a 20% improvement in response (per the Assessment in Ankylosing Spondylitis International Working Group) defined as meeting 2 criteria: 1) An improvement of >=20% from Baseline and an absolute improvement from Baseline of >=10 mm in at least 3 of 4 domains, and 2) Absence of deterioration from Baseline (defined as a >=20% worsening and an absolute worsening of >=10 mm) in the potential remaining domain. The percentages of participants who achieved ASAS 20 were calculated.
Time Frame: Week 16
Population: The Full-Analysis-Set (FAS) population consisted of all randomized participants who received at least one dose of study drug in Part 1.
Measure: Number; unit: Percentage of Participants
Arm/Group | Golimumab→Golimumab | Placebo→Golimumab
Number analyzed (Participants) | 97 | 100
Percentage of Participants | 71.1 | 40.0
Statistical Analysis 1: Comparison: Golimumab→Golimumab vs Placebo→Golimumab; Test type: Superiority or Other; p < 0.0001, Stratified Miettinen and Nurminen Method — Stratification factors: Baseline evidence of sacroiliitis on magnetic resonance imaging (MRI) and Screening C-reactive protein (CRP) level; Difference in Percent vs Placebo = 31.2, 95% CI 2-sided [17.5 to 43.6]

2. Secondary Outcome: Percentage of Participants Achieving an Assessment in Ankylosing Spondylitis (ASAS) 40 Response at Week 16
Description: The ASAS consists of 4 domains: participant global assessment, total back pain, function (BASFI), and inflammation (mean of questions 5 and 6 of BASDAI). Each domain is measured on a 100-mm VAS from 0 mm=the very best situation to 100 mm=the very worst situation, with a higher score indicating more severe impairment. ASAS 40 is a 40% improvement in response (per the Assessment in Ankylosing Spondylitis International Working Group) defined as meeting 2 criteria: 1) An improvement of >=40% from Baseline and an absolute improvement from Baseline of >=20 mm in at least 3 of 4 domains, and 2) Absence of deterioration from Baseline (defined as a >=0% worsening and an absolute worsening of >=0 mm) in the potential remaining domain. The percentages of participants who achieved ASAS 40 were calculated.
Time Frame: Week 16
Population: The FAS population consisted of all randomized participants who received at least one dose of study drug in Part 1.
Measure: Number; unit: Percentage of Participants
Arm/Group | Golimumab→Golimumab | Placebo→Golimumab
Number analyzed (Participants) | 97 | 100
Percentage of Participants | 56.7 | 23.0
Statistical Analysis 1: Comparison: Golimumab→Golimumab vs Placebo→Golimumab; Test type: Superiority or Other; p < 0.0001, Stratified Miettinen and Nurminen Method — Stratification factors: Baseline evidence of sacroiliitis on MRI and Screening CRP level; Difference in Percent vs Placebo = 33.8, 95% CI 2-sided [20.4 to 46.1]

3. Secondary Outcome: Percentage of Participants Achieving Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 50 at Week 16
Description: The BASDAI is a summary of 6 participant-assessed 100-mm VAS for a) Fatigue, b) Spinal pain (overall), c) Peripheral arthritis, d) Enthesitis, e) Qualitative morning stiffness (intensity) and f) Quantitative morning stiffness (duration). Each VAS is measured as 0=none to 100=very severe, with a higher score indicating more severe symptoms. The BASDAI score is calculated as 0.2 time (a+b+c+d+[0.5 times e+f]) and can range from 0 to 100. The BASDAI 50 is defined as improvement by at least 50% from Baseline in the BASDAI score. The percentages of participants who achieved BASDAI 50 were calculated.
Time Frame: Week 16
Population: The FAS population consisted of all randomized participants who received at least one dose of study drug in Part 1 and had a Baseline BASDAI assessement.
Measure: Number; unit: Percentage of Participants
Arm/Group | Golimumab→Golimumab | Placebo→Golimumab
Number analyzed (Participants) | 97 | 100
Percentage of Participants | 57.7 | 30.0
Statistical Analysis 1: Comparison: Golimumab→Golimumab vs Placebo→Golimumab; Test type: Superiority or Other; p < 0.0001, Stratified Miettinen and Nurminen Method — Stratification factors: Baseline evidence of sacroiliitis on MRI and Screening CRP level; Difference in Percent vs Placebo = 28.0, 95% CI 2-sided [14.4 to 40.6]

4. Secondary Outcome: Percentage of Participants Achieving ASAS Partial Remission at Week 16
Description: ASAS partial remission was defined as a VAS score of less than 20 mm in each of the 4 domains of ASAS 20: participant global assessment, pain (total back pain), function and inflammation. The percentages of participants who achieved ASAS partial remission were calculated.
Time Frame: Week 16
Population: The FAS population consisted of all randomized participants who received at least one dose of study drug in Part 1.
Measure: Number; unit: Percentage of Participants
Arm/Group | Golimumab→Golimumab | Placebo→Golimumab
Number analyzed (Participants) | 97 | 100
Percentage of Participants | 33.0 | 18.0
Statistical Analysis 1: Comparison: Golimumab→Golimumab vs Placebo→Golimumab; Test type: Superiority or Other; p = 0.0136, Stratified Miettinen and Nurminen Method — Stratification factors: Baseline evidence of sacroiliitis on MRI and Screening CRP level; Difference in Percent vs Placebo = 15.2, 95% CI 2-sided [3.2 to 27.1]

5. Secondary Outcome: Change From Baseline in Spondyloarthritis Research Consortium of Canada (SPARCC) Magnetic Resonance Imaging (MRI) Sacroiliac (SI) Joints Score at Week 16
Description: Participants underwent MRI of the SI joints, without contrast, at Screening and Week 16 to assess the presence or absence of active inflammation of the SI joints. Scoring was based on 6 consecutive MRI slices through the SI joint. Each slice was divided into 4 quadrants. Each of the 48 quadrants was scored with respect to the presence of inflammation (0=no, 1=yes), yielding a maximum score of 48. Each slice was also assessed for the presence of a lesion exhibiting either intense signal or a depth >=1 cm anywhere within the SI joint of the 6 slices (0=no, 1=yes), yielding a maximum score of 24. Total SI joint scores could range from 0 to 72, with a higher score indicating more signs of disease.
Time Frame: Baseline and Week 16
Population: The FAS population consisted of all randomized participants who received at least one dose of study drug in Part 1, who completed Part 1, and who had Baseline and Week 16 MRI SI joint measurements.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Golimumab→Golimumab | Placebo→Golimumab
Number analyzed (Participants) | 74 | 87
Score on a Scale
  Baseline Score | 9.87 (11.822) | 12.66 (15.619)
  Change from Baseline at Week 16 | -5.25 (7.708) | -0.95 (8.533)
Statistical Analysis 1: Comparison: Golimumab→Golimumab vs Placebo→Golimumab; Test type: Superiority or Other; p < 0.0001, Mann-Whitney Test

6. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event (AE)
Description: An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug, whether or not considered related to the study drug. The percentages of participants who experienced at least one AE were calculated for each part of the study.
Time Frame: Up to 16 weeks for Part 1: Week 16 through up to 60 weeks for Part 2 (Up to 12 weeks after last dose of study drug)
Population: The All-Participants-as-Treated (APaT) population of this study consisted of all randomized participants who received at least one dose of study drug. These data are for Parts 1 and 2 of the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | Golimumab→Golimumab | Placebo→Golimumab
Number analyzed (Participants) | 97 | 100
Percentage of Participants
  Part 1 (Up to 16 weeks) (n=97, 100) | 41.2 | 47.0
  Part 2 (Up to 60 weeks) (n=93, 96) | 41.9 | 54.2

7. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an AE
Description: An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug, whether or not considered related to the study drug. The percentages of participants who discontinued study drug due to an AE were calculated for each part of the study. Participants may have discontinued study drug without discontinuing from the study.
Time Frame: Up to 16 weeks for Part 1; Week 16 through up to 48 weeks for Part 2
Population: The APaT population of this study consisted of all randomized participants who received at least one dose of study drug. These data are for Parts 1 and 2 of the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | Golimumab→Golimumab | Placebo→Golimumab
Number analyzed (Participants) | 97 | 100
Percentage of Participants
  Part 1 (Up to 16 weeks) (n=97, 100) | 2.1 | 1.0
  Part 2 (Up to 52 weeks) (n=93, 96) | 1.1 | 2.1

ADVERSE EVENTS:
Time Frame: Up to 16 weeks for Part 1: Week 16 through up to 60 weeks for Part 2 (Up to 12 weeks after last dose of study drug)
Description: The All-Participants-as-Treated (APaT) population of this study consisted of all randomized participants who received at least one dose of study drug. These data are for Parts 1 and 2 of the study.
Groups:
- Part 1: Golimumab→Golimumab; Part 2: Golimumab→Golimumab: In Part 1, participants receive golimumab 50 mg, administered SC every 4 weeks for up to 12 weeks (16 weeks of treatment). In Part 2, participants receive golimumab 50 mg, administered SC every 4 weeks for up to 28 weeks (32 weeks of treatment). (Combined total of up to 48 weeks treatment with golimumab.)
- Part 1: Placebo→Golimumab; Part 2: Placebo→Golimumab: In Part 1, participants receive placebo, administered SC every 4 weeks for up to 12 weeks (16 weeks of treatment). In Part 2, participants receive golimumab 50 mg, administered SC every 4 weeks for up to 28 weeks (32 weeks of treatment). (Combined total of up to 32 weeks treatment with golimumab.)
Arm/Group | Part 1: Golimumab→Golimumab | Part 1: Placebo→Golimumab | Part 2: Golimumab→Golimumab | Part 2: Placebo→Golimumab
Serious Adverse Events (participants affected / at risk) | 1/97 | 2/100 | 2/93 | 3/96
Other Adverse Events (participants affected / at risk) | 17/97 | 21/100 | 13/93 | 27/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Golimumab→Golimumab (N=97) | Part 1: Placebo→Golimumab (N=100) | Part 2: Golimumab→Golimumab (N=93) | Part 2: Placebo→Golimumab (N=96)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Golimumab→Golimumab (N=97) | Part 1: Placebo→Golimumab (N=100) | Part 2: Golimumab→Golimumab (N=93) | Part 2: Placebo→Golimumab (N=96)
Nausea (Gastrointestinal disorders) | 0 (0) | 6 (8) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 9 (11) | 9 (11) | 5 (5) | 10 (12)
Headache (Nervous system disorders) | 7 (8) | 6 (11) | 6 (11) | 8 (26)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (5) | 6 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the study without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication (including slides and texts of oral or other public presentations and texts of any transmission through any electronic media) that report any results of the trial.